CLINICAL TRIAL: NCT05247944
Title: Propensity Matched Comparison of Fenestrated Endovascular Aneurysm Repair and Open Surgical Repair for Complex Abdominal Aortic Aneurysms.
Brief Title: F-BEVAR vs Open Surgery for Complex Abdominal Aortic Aneurysm
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Head of the Endovascular Therapies Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1843
Record Dates: First submitted 2022-01-31; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Aneurysm Aortic; Vascular Diseases
Keywords: F-BEVAR; Open surgery; complex abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- F-BEVAR: Patients with complex abdominal aortic aneurysm who underwent fenestrated and branched endovascular aortic repair (F-BEVAR) at the Aortic Center of Lille (ACL; Lille, France).
  Interventions: Procedure: Fenestrated and branched endovascular aortic repair (F-BEVAR)
- OPEN SURGERY REPAIR: Patients with complex abdominal aortic aneurysm who underwent open surgery repair the Unit of Vascular Surgery of Policlinic Gemelli (FPUG; Rome, Italy).
  Interventions: Procedure: Open repair

INTERVENTIONS:
Procedure: Fenestrated and branched endovascular aortic repair (F-BEVAR) — Fenestrated and branched endovascular aortic repair (F-BEVAR)
  Groups: F-BEVAR
Procedure: Open repair — Open surgery for complex abdominal aortic aneurysm
  Groups: OPEN SURGERY REPAIR

SUMMARY:
The aim of the present study was to investigate outcomes of a propensity matched series of patients treated with F-BEVAR and open surgery repair for complex abdominal aortic aneurysm in two aortic high-volume centres.

DETAILED DESCRIPTION:
This retrospective study analyzes the long-term outcomes of a propensity-matched cohort of patients with complex abdominal aortic aneurysm prospectively collected between January 2010 and June 2016 from the Aortic Center of Lille (Lille, France) and the Unit of Vascular Surgery of Policlinic Gemelli (Rome, Italy).

Patients were observed with regular postoperative appointments. The long-term imaging follow-up consisted in a yearly computed tomography angiography in the F-BEVAR group; and yearly abdominal ultrasound examination and 5-year computed tomography angiography were performed in the open surgery repair group. In case of abnormal renal function (eGFR<60 mL/min/1.73 m2), the patient underwent computed tomography without contrast associated to a contrast-enhanced ultrasound examination in both groups. Laboratory data with evaluation of renal function by estimated glomerular filtration rate (eGFR), were completed at three, six, and 12 months, and yearly thereafter. Survival assessment was completed after general partitioner's, patients' or patient siblings' contact by phone.

ELIGIBILITY:
Inclusion Criteria:

* juxtarenal abdominal aortic aneurysms
* pararenal abdominal aortic aneurysms
* suprarenal abdominal aortic aneurysms
* type IV thoracoabdominal aneurysms

Exclusion Criteria:

* extent I to III thoracoabdominal aneurysms
* ruptured o symptomatic aneurysms
* dissections or connective tissue disorder aneurysms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 157 patients, referred to the Aortic Center of Lille (France), underwent F-BEVAR treatment; 119 patients, referred to the Policlinic Gemelli in Rome (Italy), concurrently underwent OSR.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2010-01; Primary Completion 2018-01-31 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Overall mortality | Through study completion, an average of 5 year
  All cause death
Aortic-related mortality | Through study completion, an average of 5 year
  Any death related to the initial procedure.
Chronic renal decline during follow-up | Through study completion, an average of 5 year
  Chronic renal decline was defined in patients with normal (stage 1-2) preoperative renal function as a reduction in the eGFR to <60 mL/min/1.73 m2 during follow-up. In patients with abnormal function (stages 3 and 4) preoperatively, it was defined as an eGFR reduction of >20% or de novo dependence on permanent renal replacement therapy.

SECONDARY OUTCOMES:
Aortic-related reintervention | Through study completion, an average of 5 year
  All secondary interventions related to the initial procedure or to the endograft and its target vessels during follow-up
Target vessel occlusion | Through study completion, an average of 5 year
  Complete obstruction of the artery with no evidence of flow identified on any follow-up CT scan or duplex ultrasound.
Clinical failure | Through study completion, an average of 5 year
  Death from complications of the initial operation or a secondary intervention, aortic aneurysm rupture, aortic conversion to open surgical repair, persistent type I or III endoleak, sac expansion >5 mm, device migration >10mm, infection or thrombosis in the F-BEVAR group and death, graft infection or thrombosis or para-anastomotic aneurysm in the open group.
Proximal aorta degeneration Proximal aorta degeneration | Through study completion, an average of 5 year
  Diameter increase >5 mm within 5 cm above the ostium of the more proximal target vessel for the endovascular group and 5 cm above the proximal anastomosis for the open group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinelli G, Crea MA, de Waure C, Di Tanna GL, Becquemin JP, Sobocinski J, Snider F, Haulon S. A propensity-matched comparison of fenestrated endovascular aneurysm repair and open surgical repair of pararenal and paravisceral aortic aneurysms. J Vasc Surg. 2018 Sep;68(3):659-668. doi: 10.1016/j.jvs.2017.12.060. Epub 2018 Mar 22. PMID 29576405